CLINICAL TRIAL: NCT03960502
Title: A Phase I, Open-label Study to Evaluate the Absorption, Distribution, Metabolism, and Excretion, and to Assess the Absolute Bioavailability of AG-881 in Healthy Male Subjects Following Administration of a Single Oral Dose of [14C] AG-881 and Concomitant Intravenous Microdose of [13C315N3] AG-881
Brief Title: A Safety and Pharmacokinetic Study of AG-881 in Healthy Male Participants Following Administration of a Single Oral Dose of [14C] AG-881 and Concomitant Intravenous Microdose of [13C315N3] AG-881
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Agios Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: AG881-C-005
Record Dates: First submitted 2019-05-21; First posted 2019-05-23 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Healthy Male Participants
Keywords: Safety and tolerability; Pharmacokinetic study

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AG881 (Experimental): On Day 1, after fasting for 10 hours participants, will receive an oral capsule of [14C]AG-881 followed 2 hours later by a single intravenous (IV) infusion of [13C315N3]AG-881.
  Interventions: Drug: AG-881; Drug: [13C315N3]AG-881

INTERVENTIONS:
Drug: AG-881 — Single oral dose of approximately 50 mg AG-881 (free form) containing approximately 100 microcuries (μCi) of [14C]AG-881.
Drug: [13C315N3]AG-881 — Single IV microdose of approximately 100 μg.

SUMMARY:
The purpose of this Phase I, open-label study is to evaluate the absorption, distribution, metabolism, excretion, absolute bioavailability, and to characterize the metabolites of AG-881 in healthy male participants following administration of a single oral dose of [14C] AG-881 and a concomitant intravenous microdose of [13C315N3] AG-881.

ELIGIBILITY:
Inclusion Criteria:

* Able to comprehend and willing to sign an informed consent form (ICF) and to abide by the study restrictions, including confinement, as well as adhere to all study procedures;
* Males of any race, between 18 and 55 years of age, inclusive;
* Body mass index between 18.0 and 32.0 kilograms per meter squared (kg/m^2), inclusive, and a total body weight between 50 and 100 kg, inclusive;
* In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead electrocardiogram (ECG), vital sign measurements, and clinical laboratory evaluations (congenital non-hemolytic hyperbilirubinemia [e.g., suspicion of Gilbert's syndrome based on total and direct bilirubin] is not acceptable) at Screening and/or Check-in (Day -1), as assessed by the Investigator (or designee);
* Alanine aminotransferase (ALT; at or within normal limits [WNL]), aspartate aminotransferase (AST; at or within normal limits), alkaline phosphatase (ALP; <1.5 × upper limit of normal [ULN]), bilirubin (at or below WNL). One repeat assessment allowed at each time point;
* Male participants will agree to use contraception;
* Agrees to abstain from any alcohol consumption, starting 48 hours before Check-in (Day -1) and continuing until Discharge;
* History of a minimum of one bowel movement per day;
* Adequate peripheral venous access.

Exclusion Criteria:

* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the Investigator (or designee);
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator (or designee);
* History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (uncomplicated appendectomy and hernia repair will be allowed);
* Has undergone any major surgical procedure within the 3 months prior to Screening;
* History of alcoholism or drug/chemical abuse within 2 years prior to Check-in (Day -1);
* History of severe and/or uncontrolled ventricular arrhythmias or other factors that increase the risk of long QT syndrome, or use, or intend to use, medications that are known to prolong the QT interval or history of unexplained syncopal events or familial history of unexplained death in young person;
* After at least 5 minutes of rest in the supine position at Screening, has a systolic blood pressure reading of ≥140 millimeters of mercury (mmHg) OR a diastolic blood pressure reading of ≥90 mmHg;
* A heart rate-corrected QT interval by Fridericia's (QTcF) method of ≥450 milliseconds (ms);
* Alcohol consumption of >21 units per week. One unit of alcohol equals 12 ounces (360 millimeters [mL]) of beer, 1½ oz (45 mL) of liquor, or 5 oz (150 mL) of wine;
* Positive urine drug screen at Screening or positive alcohol breath test result or positive urine drug screen at Check-in (Day -1);
* Positive hepatitis panel and/or positive human immunodeficiency virus test;
* Participation in a clinical study involving administration of an investigational drug (new chemical entity) in the past 30 days or 5 half-lives (whichever is longer), prior to dosing;
* Use or intend to use any medications/products known to alter drug absorption, metabolism, or elimination processes, including St. John's wort, within 30 days prior to Check-in (Day -1), unless deemed acceptable by the Investigator (or designee);
* Use or intend to use any prescription medications/products within 14 days prior to Check-in (Day -1), unless deemed acceptable by the Investigator (or designee);
* Use or intend to use slow-release medications/products considered to still be active within 30 days prior to Check-in (Day -1), unless deemed acceptable by the Investigator (or designee);
* Use or intend to use any nonprescription medications/products including vitamins, minerals, and phytotherapeutic/herbal/plant-derived preparations within 7 days prior to Check-in (Day -1), unless deemed acceptable by the Investigator (or designee);
* Use of tobacco- or nicotine-containing products within 3 months prior to Check-in (Day -1), or positive cotinine at Screening or Check-in (Day -1);
* Receipt of blood products within 2 months prior to Check-in (Day -1);
* Donation of blood from 3 months prior to Screening, plasma from 2 weeks prior to Screening, or platelets from 6 weeks prior to Screening;
* Have previously completed or withdrawn from this study or any other study investigating AG-881, and have previously received the investigational product;
* Participants with exposure to significant diagnostic or therapeutic radiation (e.g., serial X-ray, computed tomography scan, barium meal) or current employment in a job requiring radiation exposure monitoring within 12 months prior to Check-in (Day -1);
* Participants who have participated in a radiolabeled drug study where exposures are known to the Investigator within the previous 4 months prior to admission to the clinic for this study or participated in a radiolabeled drug study where exposures are not known to the Investigator within the previous 6 months prior to admission to the clinic for this study. The total 12-month exposure from this study and a maximum of 2 other previous radiolabeled studies within 4 to 12 months prior to this study will be within the Code of Federal Regulations (CFR) recommended levels considered safe, per United States (US) Title 21 CFR 361.1: less than 5,000 millirems (mrem) whole-body annual exposure with consideration given to the half-lives of the previous radiolabeled study drugs received;
* Is an employee of, or an immediate family member of an employee of, the study site or the Sponsor;
* Participants who, in the opinion of the Investigator (or designee), should not be part of this study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2019-05-16 (Actual); Primary Completion 2019-09-07 (Actual); Study Completion 2019-09-07 (Actual)

PRIMARY OUTCOMES:
Amount of AG-881 Excreted in Urine (Aeu) | At multiple time points daily from Day -1 to Day 14; then at 24-hour intervals until discharge (up to 29 days); then weekly up to approximately 8 weeks
Cumulative Aeu (Cum Aeu) of AG-881 | At multiple time points daily from Day -1 to Day 14; then at 24-hour intervals until discharge (up to 29 days); then weekly up to approximately 8 weeks
Percentage of AG-881 excreted in Urine and Feces (feu and fef, Respectively) | At multiple time points daily from Day -1 to Day 14; then at 24-hour intervals until discharge (up to 29 days); then weekly up to approximately 8 weeks
Cumulative Percentage of AG-881 Excreted in Urine (Cum feu) | At multiple time points daily from Day -1 to Day 14; then at 24-hour intervals until discharge (up to 29 days); then weekly up to approximately 8 weeks
Cumulative Percentage of AG-881 Excreted in Feces (Cum fef) | At multiple time points daily from Day -1 to Day 14; then at 24-hour intervals until discharge (up to 29 days); then weekly up to approximately 8 weeks
Renal Clearance (CLR) of AG-881 | At multiple time points daily from Day -1 to Day 14; then at 24-hour intervals until discharge (up to 29 days); then weekly up to approximately 8 weeks
Renal Clearance Expressed as a Percentage of Total Clearance (CLR/CL) of AG-881 | At multiple time points daily from Day -1 to Day 14; then at 24-hour intervals until discharge (up to 29 days); then weekly up to approximately 8 weeks
Percentage of Total Radioactivity in Total Excreta Calculated as Cumulative Percentage of AG-881 Excreted in Urine and Feces (Cum fe) | At multiple time points daily from Day -1 to Day 14; then at 24-hour intervals until discharge (up to 29 days); then weekly up to approximately 8 weeks
Area Under the Concentration-time Curve from Time Zero to the Last Measurable Concentration (AUC0-last) of AG-881 | At multiple time points daily from Day -1 to Day 14; then at 24-hour intervals until discharge (up to 29 days); then weekly up to approximately 8 weeks
Area Under the Concentration-time Curve from Time Zero to 72 hours (AUC0-72) of AG-881 | Up to 72 hours
Partial Area Under the Concentration-time Curve from Time Zero to Common Time Point (AUC0-t) of AG-881 | At multiple time points daily from Day -1 to Day 14; then at 24-hour intervals until discharge (up to 29 days); then weekly up to approximately 8 weeks
Area Under the Concentration-time Curve from Time Zero to Infinity (AUC0-∞) of AG-881 Calculated Using the Observed Value of the Last Quantifiable Concentration | At multiple time points daily from Day -1 to Day 14; then at 24-hour intervals until discharge (up to 29 days); then weekly up to approximately 8 weeks
Maximum Observed Plasma Concentration (Cmax) of AG-881 | At multiple time points daily from Day -1 to Day 14; then at 24-hour intervals until discharge (up to 29 days); then weekly up to approximately 8 weeks
Time to Maximum Observed Plasma Concentration (Tmax) of AG-881 | At multiple time points daily from Day -1 to Day 14; then at 24-hour intervals until discharge (up to 29 days); then weekly up to approximately 8 weeks
Apparent Terminal Elimination Half-life (t½) of AG-881 | At multiple time points daily from Day -1 to Day 14; then at 24-hour intervals until discharge (up to 29 days); then weekly up to approximately 8 weeks
AUC0-∞ or AUC0-t of AG-881 in Plasma/AUC0-∞ or AUC0-t of Total Radioactivity in Plasma (AUC Plasma AG-881/Total Radioactivity Ratio) | At multiple time points daily from Day -1 to Day 14; then at 24-hour intervals until discharge (up to 29 days); then weekly up to approximately 8 weeks
AUC0-∞ of Total Radioactivity in Whole Blood to AUC0-∞ of Total Radioactivity in Plasma (AUC Blood/Plasma Ratio), Calculated Using the Observed Value of the Last Quantifiable Concentration | At multiple time points daily from Day -1 to Day 14; then at 24-hour intervals until discharge (up to 29 days); then weekly up to approximately 8 weeks
Total Clearance of AG-881 Following Intravenous (IV) Administration (CL) | At multiple time points daily from Day -1 to Day 14; then at 24-hour intervals until discharge (up to 29 days); then weekly up to approximately 8 weeks
Apparent Clearance Following Oral Administration of AG-881 (CL/F) | At multiple time points daily from Day -1 to Day 14; then at 24-hour intervals until discharge (up to 29 days); then weekly up to approximately 8 weeks
Volume of Distribution of AG-881 at Steady-state Following IV Administration (Vss) | At multiple time points daily from Day -1 to Day 14; then at 24-hour intervals until discharge (up to 29 days); then weekly up to approximately 8 weeks
Apparent Volume of Distribution During the Terminal Phase Following Oral Administration of AG-881 (Vz/F) | At multiple time points daily from Day -1 to Day 14; then at 24-hour intervals until discharge (up to 29 days); then weekly up to approximately 8 weeks
Absolute bioavailability (F) for AG-881 Calculated as the Ratio of Dose-normalized AUC0-∞ of Oral/Intravenous Dosing | At multiple time points daily from Day -1 to Day 14; then at 24-hour intervals until discharge (up to 29 days); then weekly up to approximately 8 weeks
Metabolic Profiles of AG-881 in Plasma, Urine, and Feces, When Possible | At multiple time points daily from Day -1 to Day 14; then at 24-hour intervals until discharge (up to 29 days); then weekly up to approximately 8 weeks
Structures of AG-881 Metabolites in Plasma, Urine, and, Where Possible, Feces | At multiple time points daily from Day -1 to Day 14; then at 24-hour intervals until discharge (up to 29 days); then weekly up to approximately 8 weeks

SECONDARY OUTCOMES:
Percentage of Participants with Adverse Events (AEs), Graded by Severity | Up to approximately 12 weeks
  AEs will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE; Version 4.03)
Percentage of Participants with Laboratory Abnormalities | Up to approximately 8 weeks
  Laboratory assessments will include parameters assessing clinical chemistry, hematology, coagulation, urinalysis, and serology.
Percentage of Participants with Abnormalities in 12-lead Electrocardiogram (ECG) | Up to approximately 8 weeks
Percentage of Participants with Abnormalities in Vital Signs Measurements | Up to approximately 8 weeks
  Vital signs will include supine blood pressure, supine pulse rate, and oral body temperature.
Percentage of Participants with Abnormalities in Physical Examinations | Up to approximately 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Affairs, Study Chair — Agios Pharmaceuticals, Inc.
Locations (1):
- Covance Clinical Research Unit Inc., Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No